CLINICAL TRIAL: NCT05437302
Title: Effectiveness of Prism Spectacles in Patients With Age Related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, mehreen tanveer, principal investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ufaisalabad
Record Dates: First submitted 2022-06-10; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): prism spectacles prescribed
  Interventions: Device: prism spectacle
- non interventional (Active Comparator): presbyopia glasses prescribed
  Interventions: Device: prism spectacle

INTERVENTIONS:
Device: prism spectacle — a prism is dispensed in prescription glasses

SUMMARY:
A study is conducted to determine the effectiveness of prism spectacles in improving visual acuity with age related macular degeneration patients and to assess the improvement in quality of life in patients by using prism spectacles.

DETAILED DESCRIPTION:
A random sampling technique will be used to allocate patient in interventional and non-interventional group. The diagnosed patients of age-related macular degeneration are assessed for prism spectacles for near vision and prism glasses will be dispensed to the patients. Each subject will be interviewed to fill the Proforma after taking the informed consent. The results of this study will show the effectiveness of prism glasses in patients with age related macular degeneration in their daily routine near work as compared to conventional glasses.

ELIGIBILITY:
Inclusion Criteria:

* Patients having age >50 years with age related macular degeneration.
* Patients of both genders (male and female).
* Participants who will be willing to give informed consent for participation in the study.

Exclusion Criteria:

* Presence of all ocular disease and systemic ocular pathologies able to impair visual function.
* Presence of disorders causing choroidal neovascularization other than age related macular degeneration.
* Patients with mental illness, dementia, and severe physical limitations

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | Four week
  Near and Distance visual acuity are measured in log Mar units.
Visual Functional Quality of life (VFQOL) | Four weeks
  VFQOL is measured by a validated tool VFQOL-25.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Kiran, Study Director — University of Faisalabad
Locations (1):
- Mehreen, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No